CLINICAL TRIAL: NCT01960413
Title: Phase 2 Study of Montelukast for the Treatment of Sickle Cell Anemia (Also Known as the Montelukast Trial in Sickle Cell Anemia)
Brief Title: Phase 2 Study of Montelukast for the Treatment of Sickle Cell Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Medical College of Wisconsin (Other); Versiti Blood Health (Other)
Responsible Party: Principal Investigator, Michael DeBaun, Professor of Pediatrics and Medicine, JC Peterson Endowed Chair in Pediatrics, Vice Chair for Clinical Research in Pediatrics, Director, Vanderbilt-Meharry-Matthew Walker Center for Excellence in Sickle Cell Disease, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R01FD004117 (FDA)
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Results first posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Sickle Cell Anemia (HbSS, or HbSβ-thalassemia0)
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Montelukast added to Hydroxyurea (Experimental): Oral montelukast therapy taken daily for eight weeks with current hydroxyurea regiment
  Interventions: Drug: Montelukast added to Hydroxyurea
- Placebo added to Hydroxyurea (Placebo Comparator): Oral placebo taken daily for eight weeks with current hydroxyurea regiment
  Interventions: Drug: Placebo added to Hydroxyurea

INTERVENTIONS:
Drug: Montelukast added to Hydroxyurea
  Arms: Montelukast added to Hydroxyurea
Drug: Placebo added to Hydroxyurea
  Arms: Placebo added to Hydroxyurea

SUMMARY:
In this feasibility trial, the investigators will compare participants treated with montelukast and hydroxyurea to those treated with placebo and hydroxyurea for a total of 8 weeks.

DETAILED DESCRIPTION:
The primary hypothesis for this trial is that montelukast adds efficacy to hydroxyurea therapy for improving vaso-occlusion when compared to hydroxyurea alone. The following specific aims will be tested in adolescents and adults with sickle cell disease (SCD):

Aim 1. To determine whether montelukast versus placebo added to hydroxyurea will improve markers of vaso-occlusion-associated tissue injury in adolescents and adults with sickle cell disease.

Aim 2. To evaluate physiologic effects of montelukast versus placebo added to hydroxyurea in adolescents and adults with sickle cell disease.

Subaim 2A. To determine if montelukast versus placebo added to hydroxyurea will improve lung function in adolescents and adults with sickle cell disease.

Subaim 2B. To determine if montelukast versus placebo added to hydroxyurea will improve forearm microvascular blood flow in adolescents and adults with sickle cell disease, respectively.

Funding Source - FDA OOPD

ELIGIBILITY:
Inclusion Criteria:

* 1)Diagnosis of HbSS, or HbSβ-thalassemia0, confirmed by hemoglobin analysis
* 2)Males and females age 16 years to 70 years old
* 3)Greater than 2 episodes of pain in the last 12 months
* 4)On a stable dose of hydroxyurea for at least 2 months and a stable hemoglobin

Exclusion Criteria:

1. Judged not likely to be study compliant by his/her hematologist
2. History of adverse reaction to montelukast or any of the components of montelukast
3. Have used medications known to interact with montelukast such as rifampin, phenobarbital, and gemfibrozil within 4 weeks of enrollment
4. Currently being treated with a leukotriene antagonist (montelukast or zileuton) or have used montelukast/zileuton within the last 60 days
5. Chronic blood transfusion therapy defined as regularly scheduled transfusions.
6. Hemoglobin A greater than15% on hemoglobin analysis
7. Individuals with a current physician diagnosis of asthma (within last 12 months) or requires continuous supplemental oxygen, or predicted or current use of asthma medications (inhaled corticosteroids, but participants taking bronchodilators will be allowed to participate).
8. Current participation in another therapeutic trial for SCD
9. Known current pregnancy
10. Known history of HIV
11. Serum creatinine greater than 3 times the site's upper limit of normal

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2013-11; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael R. DeBaun, MD, MPH, Principal Investigator — Vanderbilt University Medical Center; Joshua Field, MD, MS, Principal Investigator — Medical College of Wisconsin
Locations (2):
- United States (2):
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identiﬁcation (text, tables, ﬁgures, and appendices)
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.

REFERENCES:
- [Derived] Field JJ, Kassim A, Brandow A, Embury SH, Matsui N, Wilkerson K, Bryant V, Zhang L, Simpson P, DeBaun MR. Phase 2 trial of montelukast for prevention of pain in sickle cell disease. Blood Adv. 2020 Mar 24;4(6):1159-1165. doi: 10.1182/bloodadvances.2019001165. PMID 32208487

RESULTS

PARTICIPANT FLOW:
Groups:
- Montelukast Added to Hydroxyurea: Oral montelukast therapy taken daily for eight weeks with current hydroxyurea regiment
  Montelukast added to Hydroxyurea
- Placebo Added to Hydroxyurea: Oral placebo taken daily for eight weeks with current hydroxyurea regiment
  Placebo added to Hydroxyurea
Period: Overall Study
Arm/Group | Montelukast Added to Hydroxyurea | Placebo Added to Hydroxyurea
Started | 24 | 22
Completed | 20 | 21
Not Completed | 4 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Montelukast Added to Hydroxyurea | Placebo Added to Hydroxyurea | Total
Number analyzed (Participants) | 24 | 22 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.25 (10.46) | 30.76 (10.24) | 29.95 (10.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 11 | 8 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 23 | 22 | 45
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 24 | 18 | 42
  White | 0 | 1 | 1
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 22 | 46

OUTCOME MEASURES:

1. Primary Outcome: Change in Soluble Vascular Cell Adhesion Molecule-1 (sVCAM)
Description: The primary outcome measure is based on a 30% reduction, which would be ~106 ng/ml reduction. The study was designed with 25 in each group in order to explore all three aims and potential confounders. However, if the investigators are not able to accrue 25 subjects in each arm, the investigators would still be able to detect a 30% difference in sVCAM with 17 subjects in each group. The 95% confidence interval for detecting a 30% difference is between 204 ng/ml and 290 ng/ml (or an 18-42% reduction in sVCAM). Importantly, the lower limit of the 95% confidence interval (18%) is still a clinically relevant reduction in sVCAM. Thus, if the investigators detect a 30% or larger difference in sVCAM in this study, the investigators will be assured that, based on the 95% confidence interval, these data are clinically important.
Time Frame: baseline to eight weeks
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Montelukast Added to Hydroxyurea | Placebo Added to Hydroxyurea
Number analyzed (Participants) | 20 | 21
ng/mL | -3.2 [-13.6 to 11.6] | 4.17 [-3.3 to 12.1]

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Montelukast Added to Hydroxyurea | Placebo Added to Hydroxyurea
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/22
Serious Adverse Events (participants affected / at risk) | 4/24 | 2/22
Other Adverse Events (participants affected / at risk) | 10/24 | 12/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Montelukast Added to Hydroxyurea (N=24) | Placebo Added to Hydroxyurea (N=22)
Pain (Blood and lymphatic system disorders) | 2 (2) | 2 (2) — Sickle Cell Pain Crisis/Acute Chest Syndrome
Acute Chest Syndrome (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Montelukast Added to Hydroxyurea (N=24) | Placebo Added to Hydroxyurea (N=22)
Pain (Blood and lymphatic system disorders) | 3 (4) | 6 (9)
diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (3)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
headache (General disorders) | 0 | 1 (1)
ear injury (Ear and labyrinth disorders) | 0 | 1 (2)
scleral disorder (Eye disorders) | 1 (1) | 0 (0)
headache, migraine (Nervous system disorders) | 0 (0) | 1 (2)
vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0)
urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0)
pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
flu like symptoms (Infections and infestations) | 0 (0) | 0 (0)
stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
penile pain/priapsm (Reproductive system and breast disorders) | 1 (1) | 1 (1)
sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
pain,dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
systolic murmur (Cardiac disorders) | 1 (1) | 0 (0)
Breast Infection (Infections and infestations) | 0 (0) | 1 (1)
Injury,laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pain (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-10): https://cdn.clinicaltrials.gov/large-docs/13/NCT01960413/Prot_SAP_000.pdf